CLINICAL TRIAL: NCT04054765
Title: A Virtual Reality Videogame for E-cigarette Prevention in Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000025177
Record Dates: First submitted 2019-08-08; First posted 2019-08-13 (Actual); Results first posted 2021-06-18 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: E-Cig Use; Vaping
Keywords: prevention; intervention
MeSH Terms: conditions — Vaping | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: non-equivalent control groups design with 285 teens ages 12-15 comparing the Invite Only VR intervention vs. treatment as usual
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teens in the Invite Only VR videogame (Experimental): 155 adolescents playing the Invite Only VR intervention
  Interventions: Device: videogame
- Teens receive treatment as usual (Other): 132 adolescents receive treatment as usual, which includes regular instruction in health class regarding the dangers of e-cigarettes
  Interventions: Other: treatment as usual

INTERVENTIONS:
Device: videogame — Invite Only VR videogame
  Arms: Teens in the Invite Only VR videogame
Other: treatment as usual — treatment as usual
  Arms: Teens receive treatment as usual

SUMMARY:
The use of the Invite Only VR, with the aim to prevent the initiation of e-cigarette use in teens by increasing their knowledge, decreasing their intentions to use e-cigarettes, influencing their harm perceptions and attitudes associated with e-cigarettes, and increasing self-efficacy associated with refusing peers involving e-cigarettes.

DETAILED DESCRIPTION:
Specific Aim #1: DEVELOPMENT: The researcher will update our current VR prototype into a polished videogame intervention using input from 4 focus groups of 5 adolescents each (n = 20), aged 12-17 and the extant literature. These focus groups will inform the development of the VR videogame intervention, Invite Only VR, for e-cigarette prevention among teens.

Specific Aim #2: EVALUATION: Conduct a pilot non-randomized cluster trial with 295 teens ages 11-14 comparing the Invite Only VR intervention vs. an attention/control non-health-related VR videogame, collecting assessment data at baseline, post-gameplay, three months and six months to determine:

1. the preliminary impact of the intervention on e-cigarette use behaviors, knowledge, nicotine addiction knowledge, perceived addictiveness of e-cigarettes, perceived likelihood of using e-cigarettes, perceptions of harm, self-efficacy to refuse, social approval of e-cigarettes, and e-cigarette social perceptions
2. the intervention's acceptability and feasibility by collecting quantitative and qualitative data on teens' satisfaction and gameplay experience of the intervention.
3. preliminary evidence of the impact of Invite Only VR on players' perception and experience of social pressure and social norm development

ELIGIBILITY:
Inclusion Criteria:

* Willing to wear a VR headset and play a video game for 45-60 minutes for 2-3 sessions and answer questions before and after playing the videogame.
* Be enrolled in Milford Middle School District

Exclusion Criteria:

* If subject does not fit the criteria above

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 287 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Hieftje, PhD, Principal Investigator — Yale University
Locations (1):
- Milford School District, Milford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 844 teens in Milford Schools met eligibility requirements. 557 were excluded for failure to provide signed parental consent for inclusion in the study
Groups:
- Teens in the Invite Only VR Videogame: 155 adolescents played the Invite Only VR intervention for 2-4 sessions for approximately 40 minutes per session. These 2-4 play sessions play took place following the pre-test at baseline. The post-test was administered immediately after the final play session.
  videogame: Invite Only VR videogame Invite Only VR is a VR, story-based videogame intervention that teaches adolescents aged 11 to 17 years about the health risks of using e-cigarettes while providing a virtual environment to practice refusing peer pressure to vape e-cigarettes.
- Teens Receive Treatment as Usual: 132 adolescents receive treatment as usual
  This includes attending regular health class in public school in which the dangers of e-cigarettes are discussed.
  treatment as usual: treatment as usual
Period: Baseline
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Started | 155 | 132
Completed | 150 | 129
Not Completed | 5 | 3
Not completed — Withdrawal by Subject | 5 | 3
Period: Post-Gameplay / 1-week Follow up
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Started | 150 | 129
Completed | 142 | 126
Not Completed | 8 | 3
Not completed — Withdrawal by Subject | 8 | 3
Period: 3-month Follow up
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Started | 142 | 126
Completed | 142 | 123
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 3
Period: 6-month Follow up
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Started | 142 | 123
Completed | 110 | 91
Not Completed | 32 | 32
Not completed — Lost to Follow-up | 32 | 32

BASELINE CHARACTERISTICS:
Groups:
- Teens Receive Treatment as Usual: 132 adolescents receive treatment as usual
  treatment as usual: treatment as usual
- Total: Total of all reporting groups
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual | Total
Number analyzed (Participants) | 155 | 132 | 287
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 155 | 132 | 287
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.4 (.56) | 12.5 (.59) | 12.45 (.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 49 | 130
  Male | 74 | 83 | 157
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 12 | 17 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 109 | 90 | 199
  More than one race | 9 | 8 | 17
  Unknown or Not Reported | 11 | 6 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 155 | 132 | 287
Current e-cigarette/JUUL user (Y/N) [Count of Participants; unit: Participants] — Participants were asked "Have you ever vaped or JUULed, even one or two hits?" Response options were "Yes" or "No."
  Participants | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants Who Report E-cigarette Use at 6 Months
Description: The researcher will measure the percent of individuals who, after playing Invite Only VR, report the initiation of e-cigarette use in comparison to the control condition.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
Participants | 0 | 0

2. Secondary Outcome: Attitudes Towards E-cigarettes Pre-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' attitudes involving e-cigarette use - pretest survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then play the videogame intervention. The survey includes 4 questions adapted from the National Youth Tobacco Survey (2014) focus on attitudes about e-cigarettes. Questions have 4 response choices ranging from 1 (strongly disagree) to 4 (strongly agree) or 1 (definitely yes) to 4 (definitely not), or 1 (very unlikely) to 4 (very likely). Some items were reverse coded so that scores of 1 always represented less healthy attitudes and scores of 4 corresponded to more healthy attitudes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating healthier attitudes.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 129
units on a scale | 3.38 (.46) | 3.21 (.54)

3. Secondary Outcome: Attitudes Towards E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' attitudes involving e-cigarette use - post-test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software) after playing the videogame intervention. The survey includes 4 questions adapted from the National Youth Tobacco Survey (2014) focus on attitudes about e-cigarettes. Questions have 4 response choices ranging from 1 (strongly disagree) to 4 (strongly agree) or 1 (definitely yes) to 4 (definitely not), or 1 (very unlikely) to 4 (very likely). Questions are reverse coded such that higher scores represent healthier attitudes towards e-cigarettes.
Time Frame: immediately after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 126
units on a scale | 3.37 (.49) | 3.24 (.54)

4. Secondary Outcome: Attitudes Towards E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' attitudes involving e-cigarette use - 3 months post-test survey. The survey includes 4 questions adapted from the National Youth Tobacco Survey (2014) focus on attitudes about e-cigarettes. Questions have 4 response choices ranging from 1 (strongly disagree) to 4 (strongly agree) or 1 (definitely yes) to 4 (definitely not), or 1 (very unlikely) to 4 (very likely). Some items were reverse coded so that scores of 1 always represented less healthy attitudes and scores of 4 corresponded to more healthy attitudes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating healthier attitudes.
Time Frame: 3 months after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 123
units on a scale | 3.36 (.5) | 3.28 (.55)

5. Secondary Outcome: Attitudes Towards E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' attitudes involving e-cigarette use - 6 months post-test survey. Participants will complete a survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 4 questions adapted from the National Youth Tobacco Survey (2014) focus on attitudes about e-cigarettes. Questions have 4 response choices ranging from 1 (strongly disagree) to 4 (strongly agree) or 1 (definitely yes) to 4 (definitely not), or 1 (very unlikely) to 4 (very likely). Some items were reverse coded so that scores of 1 always represented less healthy attitudes and scores of 4 corresponded to more healthy attitudes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating healthier attitudes.
Time Frame: 6 months after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
units on a scale | 3.48 (.44) | 3.28 (.58)

6. Secondary Outcome: Knowledge of E-cigarettes Pre-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' knowledge about e-cigarettes - pre-test survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software), before playing the videogame intervention. The survey includes 15 questions adapted from the National Youth Tobacco Survey (2014) focus on knowledge about e-cigarettes. For knowledge, questions have 3 response choices (True, False, and not sure). Correct answers are scored as 1, incorrect are scored as 0, and not sure responses are also scored as 0. Total scores range from 0 to 15, with higher scores indicating better performance.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 129
score on a scale | 11.29 (1.91) | 10.33 (2.57)

7. Secondary Outcome: Knowledge of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' knowledge about e-cigarettes- post-test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software), after playing the videogame intervention. The survey includes 15 questions adapted from the National Youth Tobacco Survey (2014) focus on knowledge about e-cigarettes. For knowledge, questions have 3 response choices (True, False, and not sure). Correct answers are scored as 1, incorrect are scored as 0, and not sure responses are also scored as 0. Total scores range from 0 to 15, with higher scores indicating better performance.
Time Frame: immediately after gameplay
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 126
score on a scale | 13.97 (1.27) | 10.45 (2.92)

8. Secondary Outcome: Knowledge of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' knowledge about e-cigarettes- 3 months post-test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 15 questions adapted from the National Youth Tobacco Survey (2014) focus on knowledge about e-cigarettes. For knowledge, questions have 3 response choices (True, False, and not sure). Correct answers are scored as 1, incorrect are scored as 0, and not sure responses are also scored as 0. Total scores range from 0 to 15, with higher scores indicating better performance.
Time Frame: 3 months after gameplay
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 123
score on a scale | 13.6 (1.29) | 11.17 (2.88)

9. Secondary Outcome: Knowledge of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' knowledge about e-cigarettes- 6 months post-test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 15 questions adapted from the National Youth Tobacco Survey (2014) focus on knowledge about e-cigarettes. For knowledge, questions have 3 response choices (True, False, and not sure). Correct answers are scored as 1, incorrect are scored as 0, and not sure responses are also scored as 0. Total scores range from 0 to 15, with higher scores indicating better performance.
Time Frame: 6 months after gameplay
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
score on a scale | 13.39 (1.96) | 11.02 (2.78)

10. Secondary Outcome: Intentions of E-cigarettes Pre-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' intentions involving e-cigarette use - pretest survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then play the videogame intervention. The survey includes 1 question adapted from the National Youth Tobacco Survey (2014): "Do you think you will vape or use an e-cigarette, like JUUL, in the next year?" Participants respond on a Likert scale ranging from 1 (not at all likely) to 5 (very likely).
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 129
units on a scale | 1.12 (.44) | 1.25 (.55)

11. Secondary Outcome: Intentions of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' intentions involving e-cigarette use - post test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software) after playing videogame intervention. The survey includes 1 question adapted from the National Youth Tobacco Survey (2014): "Do you think you will vape or use an e-cigarette, like JUUL, in the next year?" Participants respond on a Likert scale ranging from 1 (not at all likely) to 5 (very likely).
Time Frame: immediately after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 126
units on a scale | 1.08 (.27) | 1.26 (.51)

12. Secondary Outcome: Intentions of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' intentions involving e-cigarette use - 3 months post test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 1 question adapted from the National Youth Tobacco Survey (2014): "Do you think you will vape or use an e-cigarette, like JUUL, in the next year?" Participants respond on a Likert scale ranging from 1 (not at all likely) to 5 (very likely).
Time Frame: 3 months after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 123
units on a scale | 1.18 (.41) | 1.28 (.56)

13. Secondary Outcome: Intentions of E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' intentions involving e-cigarette use - 6 months post test survey. Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes 1 question adapted from the National Youth Tobacco Survey (2014): "Do you think you will vape or use an e-cigarette, like JUUL, in the next year?" Participants respond on a Likert scale ranging from 1 (not at all likely) to 5 (very likely).
Time Frame: 6 months after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
units on a scale | 1.11 (.32) | 1.21 (.44)

14. Secondary Outcome: Perceptions Involving E-cigarettes Pretest
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' harm perceptions involving e-cigarette use - pretest survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) before playing the videogame intervention. The survey includes 5 questions adapted from the National Youth Tobacco Survey (2014) focus on harm perceptions about e-cigarettes. Questions have 4 choices ranging from 1 (no harm) to 4 (a lot of harm). Some items are reverse coded such that higher mean scores indicate greater perceived harm of e-cigarettes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater perceived harm.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 129
units on a scale | 2.56 (.29) | 2.57 (.3)

15. Secondary Outcome: Perceptions Involving E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' harm perceptions involving e-cigarette use - post-test survey. Participants will complete the survey through a secured, data collection website (Qualtrics Data Collection Software) after playing the videogame intervention. The survey includes 5 questions adapted from the National Youth Tobacco Survey (2014) that focus on harm perceptions about e-cigarettes. Questions have 4 choices ranging from 1 (no harm) to 4 (a lot of harm). Some items are reverse coded such that higher scores indicate greater perceived harm of e-cigarettes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater perceived harm.
Time Frame: immediately after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 126
units on a scale | 2.69 (.24) | 2.56 (.35)

16. Secondary Outcome: Perceptions Involving E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' harm perceptions involving e-cigarette use - 3 month post-test survey. Participants complete a survey through a secured, data collection website (Qualtrics Data Collection Software) 3 months after playing the intervention. The survey includes 5 questions adapted from the National Youth Tobacco Survey (2014) that focus on harm perceptions of e-cigarettes. Questions have 4 choices ranging from 1 (no harm) to 4 (a lot of harm). Some items are reverse coded such that higher scores indicate greater perceived harm of e-cigarettes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater perceived harm.
Time Frame: 3 months after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 123
units on a scale | 2.65 (.19) | 2.57 (.3)

17. Secondary Outcome: Perceptions Involving E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' harm perceptions involving e-cigarette use - post-test survey. Participants completed a survey through a secured, data collection website (Qualtrics Data Collection Software) 6 months after playing the videogame intervention. The survey includes 5 questions adapted from the National Youth Tobacco Survey (2014) that focus on harm perceptions of e-cigarettes. Questions have 4 choices ranging from 1 (no harm) to 4 (a lot of harm). Some items are reverse coded such that higher scores indicate greater perceived harm of e-cigarettes. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater perceived harm.
Time Frame: 6 months after gameplay is completed
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
units on a scale | 2.64 (.2) | 2.55 (.23)

18. Secondary Outcome: Refuse E-cigarettes Pre-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' self-efficacy to refuse e-cigarettes - pretest survey. Participants will complete a pre-survey through a secured, data collection website (Qualtrics Data Collection Software) and then play the videogame intervention. The survey includes 6 questions adapted from the National Youth Tobacco Survey (2014) that focus on self-efficacy to refuse e-cigarettes. Questions are Likert scale and have 4 choices ranging from 1 (not at all sure) to 4 (definitely sure). Higher scores represent greater self-efficacy to refuse e-cigarettes across a variety of situations. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater elf-efficacy to refuse e-cigarettes.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 129
units on a scale | 3.87 (.31) | 3.73 (.62)

19. Secondary Outcome: Refuse E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' self-efficacy to refuse e-cigarettes - post-test survey. Participants will completed a post-survey through a secured, data collection website (Qualtrics Data Collection Software) immediately after playing the videogame intervention. The survey includes 6 questions adapted from the National Youth Tobacco Survey (2014) that focus on self-efficacy to refuse e-cigarettes. Questions are Likert scale and have 4 choices ranging from 1 (not at all sure) to 4 (definitely sure). Higher scores represent greater self-efficacy to refuse e-cigarettes across a variety of situations. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater elf-efficacy to refuse e-cigarettes.
Time Frame: immediately after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 126
units on a scale | 3.89 (.37) | 3.72 (.62)

20. Secondary Outcome: Refuse E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' self-efficacy to refuse e-cigarettes - 3 months post-test survey. Participants will completed a survey through a secured, data collection website (Qualtrics Data Collection Software) 3 months after playing the videogame intervention. The survey includes 6 questions adapted from the National Youth Tobacco Survey (2014) that focus on self-efficacy to refuse e-cigarettes. Questions are Likert scale and have 4 choices ranging from 1 (not at all sure) to 4 (definitely sure). Higher scores represent greater self-efficacy to refuse e-cigarettes across a variety of situations. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater elf-efficacy to refuse e-cigarettes.
Time Frame: 3 months after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 142 | 123
units on a scale | 3.9 (.24) | 3.77 (.53)

21. Secondary Outcome: Refuse E-cigarettes Post-test
Description: To determine the impact of a VR prevention videogame intervention prototype, Invite Only VR, on participants' self-efficacy to refuse e-cigarettes - 6 months post-test survey. Participants completed a survey through a secured, data collection website (Qualtrics Data Collection Software) 6 months after playing the videogame intervention. The survey includes 6 questions adapted from the National Youth Tobacco Survey (2014) that focus on self-efficacy to refuse e-cigarettes. Questions are Likert scale and have 4 choices ranging from 1 (not at all sure) to 4 (definitely sure). Higher scores represent greater self-efficacy to refuse e-cigarettes across a variety of situations. Items were averaged into a composite scale that ranged from 1 to 4, with higher scores indicating greater elf-efficacy to refuse e-cigarettes.
Time Frame: 6 months after gameplay
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 110 | 91
units on a scale | 3.9 (.23) | 3.83 (.44)

22. Other Pre Specified Outcome: Satisfaction With Gameplay Experience - Experimental Only
Description: To determine participants' satisfaction and gameplay experience - posttest survey (experimental only). Participants will complete a post-survey through a secured, data collection website (Qualtrics Data Collection Software). The survey includes questions adapted from a survey developed at the play2PREVENT Lab about gameplay satisfaction and experience. Questions have 4 choices ranging from strongly disagree to strongly agree. Some items were reverse coded prior to all items being averaged into a composite scale that ranged from 1 to 4, with higher scores representing greater satisfaction with gameplay experience.
Time Frame: immediately after gameplay
Population: Only teens in the Invite Only VR Videogame Group responded to this survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
Number analyzed (Participants) | 150 | 0
units on a scale | 3.08 (.59) |

ADVERSE EVENTS:
Time Frame: Adverse events collected throughout the duration of the study (~6 months)
Description: The study protocol included playing a videogame and responding to questions on a brief survey about e-cigarette knowledge and beliefs. Participants were not at risk for any serious adverse events at any time during the study.
Arm/Group | Teens in the Invite Only VR Videogame | Teens Receive Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/132
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/132
Other Adverse Events (participants affected / at risk) | 0/155 | 0/132

LIMITATIONS AND CAVEATS:
It is possible that if we had followed the participants beyond 6 months, group differences might have emerged. It is also possible that because of the COVID-19 pandemic and subsequent lockdown, participants in both groups had reduced access to e-cigarettes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-27): https://cdn.clinicaltrials.gov/large-docs/65/NCT04054765/Prot_SAP_001.pdf